CLINICAL TRIAL: NCT00192673
Title: PEG-asparaginase During Two Treatment Courses in the Treatment of Childhood Acute Lymphoblastic Leukemia
Brief Title: Poly(Ethylene Glycol)(PEG)-Asparaginase During Two Treatment Courses
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nordic Society for Pediatric Hematology and Oncology (Other)
Collaborators: Medac, Hamburg, Germany (Unknown); Danish Child Cancer Foundation (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2005-000658-56; 20040177; 2004-41-4276
Record Dates: First submitted 2005-09-11; First posted 2005-09-19 (Estimated); Last update posted 2009-09-30 (Estimated); Status verified 2009-09

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: Asparaginase; intramuscular administration; Silent antibodies; Childhood acute lymphoblastic leukemia; Side effects; 5-year EFS
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — pegaspargase

INTERVENTIONS:
Drug: PEG-asparaginase

SUMMARY:
The purpose of this study is

1. to determine the correct dose for intramuscular administration
2. to compare the frequency of antibody formation after intramuscular administration of native E.coli asparaginase and PEG-asparaginase during two treatment courses in the treatment of childhood lymphoblastic leukemia

DETAILED DESCRIPTION:
Asparaginase is used in the treatment of childhood lymphoblastic leukemia. Approximately 1/3 of the patients develops blocking antibodies against native E.coli asparaginase during the second exposure, so that they do not benefit from treatment and thus may have a worse prognosis.

PEG-asparaginase is less immunogenic so that fewer patients may develop antibodies during the second exposure.

There is no published study about the antibody formation after treatment of children with PEG-asparaginase during two treatment courses.

The first part of the study is a description of the pharmacokinetics of PEG-asparaginase after intramuscular administration in order to determine the correct dose.

The second part of the study is a comparison of antibody formation during two treatment courses after intramuscular administration og native E.coli asparaginase and PEG-asparaginase.

Other side effects than antibodies will be registered during treatment with PEG-asparaginase. Finally comparison of the 5-year EFS between the groups (native E.coli asparaginase and PEG-asparaginase as well as patients who have and have not developed antibodies) will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* 1-17 years
* Newly diagnosed ALL (high intensive)
* Treated according to the NOPHO-2000 protocol
* Treated at one of the Nordic pediatric oncology centers

Exclusion Criteria:

* <1 year and >18 years
* Newly diagnosed ALL other than high intensive
* Not treated according to the NOPHO-2000 protocol
* Not treated at one of the Nordic pediatric oncology centers
* Allergy to the contents
* Pancreatitis (Active or earlier)

Ages: 1 Year to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 85 (Estimated)
Dates: Start 2005-06; Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Determination of the dose that secures sufficient treatment during 14 days
Determination of the frequency of antibody formation during treatment with PEG-asparaginase during two treatment courses

SECONDARY OUTCOMES:
Comparison of 5-year EFS between groups

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Schrøder, M.D. PhD, Study Director — Department of Pediatrics, Skejby Hospital, Denmark and member of the Scientific Commmittee in NOPHO
Locations (1):
- Department of Pediatrics, Skejby Hospital, Aarhus, Aarhus N, Denmark

REFERENCES:
- [Derived] Albenberg L, Brensinger CM, Wu Q, Gilroy E, Kappelman MD, Sandler RS, Lewis JD. A Diet Low in Red and Processed Meat Does Not Reduce Rate of Crohn's Disease Flares. Gastroenterology. 2019 Jul;157(1):128-136.e5. doi: 10.1053/j.gastro.2019.03.015. Epub 2019 Mar 11. PMID 30872105